CLINICAL TRIAL: NCT01640366
Title: A Prospective, Randomized, Intra-patient, Comparative, Open, Multi-centre Study to Evaluate the Efficacy of a Single-Use NPWT System on the Prevention of Incision Healing Complications in Patients Undergoing Reduction Mammoplasty
Brief Title: PICO Breast Reduction Clinical Study Looking at Incision Healing Complications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CE/US/11/01/PIC
Record Dates: First submitted 2012-07-03; First posted 2012-07-13 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Delayed Healing
Keywords: surgical incision; reduction mammoplasty; healing complications; negative pressure wound therapy
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PICO negative pressure (Experimental): Single-use Negative Pressure Wound Therapy
  Interventions: Device: PICO
- Standard of care dressing arm (No Intervention): Sterile gauze adhesive strips

INTERVENTIONS:
Device: PICO — Single-use Negative Pressure Wound Therapy System
  Other Names: Disposable NPWT
  Arms: PICO negative pressure

SUMMARY:
The purpose of this study is to see if the use of a single-use negative pressure wound therapy system (NPWT) will have an effect on the reduction of post-surgical incision healing complications following breast reduction surgery and to assess the medium-term aesthetic appearance and quality of the resultant scar, compared with standard of care dressings.

DETAILED DESCRIPTION:
The aim of the present study is to assess the efficacy and cost-effectiveness of the Single-Use Negative Pressure Wound Therapy (NPWT) system (PICO) with regard to the reduction of postsurgical incision healing complications during the immediate postoperative treatment phase, and to assess the medium-term aesthetic appearance and quality of the resultant scar, in patients undergoing reduction mammoplasty, compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Female patient's ≥ 18 years old
* The patient is able to understand the trial and is willing to consent to the trial
* Patient has undergone an elective surgical procedure for bilateral reduction mammoplasty
* Patients postsurgical incisions are of similar length

Exclusion Criteria:

* Pregnant or lactating females
* Patients on steroids or other immune modulators known to impact healing which may affect scar appearance
* Patients with tattoos in the area of the incisions
* Patients with skin conditions (Cutis laxa etc.) that would result in poor healing or widened scars
* Patients with a known significant history of scar problems i.e. hypertrophic scaring or keloids
* Patients who in the opinion of the investigator may not complete the study for any reason
* Patients with a known history of poor compliance with medical treatment
* Patients who have participated in this trial previously and who were withdrawn
* Patients with known allergies to product components (silicone adhesives and polyurethane films (direct contact with wound), acrylic adhesives (direct contact with skin), polyethylene fabrics and super-absorbent powders (polyacrylates) (within the dressing)
* Incisions that are actively bleeding
* Exposure of blood vessels, organs, bone or tendon at the base of the reference wound
* Incisions > 12 inches (30cm) max linear dimension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Galiano, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (6):
- United States (3):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Montefiore, The Bronx, New York
  - Cleveland Clinic, Cleveland, Ohio
- CHU de Nantes Hôtel Dieu, Nantes, France
- Academisch Ziekenhuis Maastricht (AZM), Maastricht, Netherlands
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 200 participants enrolled in this study.
Groups:
- PICO Negative Pressure Wound Therapy/Standard of Care Dressing: PICO (single-use Negative Pressure Wound Therapy system [su-NPWT]) or standard of care dressing (sterile gauze adhesive strips) were randomized to either breast following bilateral breast reduction surgery for concomitant treatment to assess the aesthetic appearance and quality of resultant scar.
Period: Overall Study
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Started | 200
Day 21 Follow-up | 185
Day 42 Follow-up | 177
Day 90 Follow-up | 178
Completed | 178
Not Completed | 22
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 16
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: 200 participants were enrolled, but 1 subject never attended any follow-up visits and was thus excluded from all data.
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 199
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 66
  African American | 50
  Hispanic | 22
  Other | 55
Region of Enrollment [Number; unit: participants]
  Netherlands | 33
  United States | 91
  France | 8
  South Africa | 68
BMI [Mean (Inter-Quartile Range); unit: kg/m^2] | 30.0 [18.1 to 57.3]
Administration of Prophylactic Antibiotics [Count of Participants; unit: Participants]
  Yes | 188
  No | 11
Surgical Technique [Count of Participants; unit: Participants]
  Superior pedicle | 18
  Inferior pedicle (with inverted "T" incision) | 55
  Superior and inferior pedicle | 6
  Superior pedicle and superomedial | 2
  Other | 118
Duration of Surgery [Mean (Inter-Quartile Range); unit: minutes] | 168.3 [49 to 445]
Mean Tissue Resection Weight [Count of Participants; unit: Participants]
  < 500 g | 68
  500 - <1000 g | 82
  1000 - <1500 g | 31
  > 1500 g | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Incision Healing Complications up to Day 21 Postoperatively
Description: The primary variable of whether or not the incision developed a healing complication within 21 days of surgery was defined as the presence of at least one of the following:
  1. Infection (superficial or deep),
  2. Dehiscence (partial, superficial or deep),
  3. Delayed healing (defined as incision not closed within 7 days of the first surgical procedure).
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery.
Measure: Number; unit: participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
participants
  PICO treatment with healing complications | 113
  PICO treatment without healing complications | 86
  Standard care with healing complications | 123
  Standard care without healing complications | 76

2. Secondary Outcome: Number of Participants Experiencing Postsurgical Incision Healing Complications (Dehiscence) Occurring up to Day 21 Postoperatively
Description: Assessment of the number of participants' incisions that experienced dehiscence (superficial, partial, or deep) occurring up to and 21 days postoperatively between incisions treated with PICO compared with standard care dressings.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery. All available results at this time point.
Measure: Number; unit: participants
Groups:
- PICO Negative Pressure Wound Therapy: PICO: Single-use Negative Pressure Wound Therapy system (su-NPWT)
Arm/Group | PICO Negative Pressure Wound Therapy
Number analyzed (Participants) | 199
participants
  PICO treatment with wound dehiscence: number analyzed (Participants) | 197
  PICO treatment with wound dehiscence | 32
  PICO treatment without wound dehiscence: number analyzed (Participants) | 197
  PICO treatment without wound dehiscence | 165
  Standard care with wound dehiscence: number analyzed (Participants) | 197
  Standard care with wound dehiscence | 52
  Standard care without wound dehiscence: number analyzed (Participants) | 197
  Standard care without wound dehiscence | 145

3. Secondary Outcome: Number of Participants Experiencing Postsurgical Incision Healing Complications (Infection) Occurring up to Day 21 Postoperatively
Description: Assessment of the number of participants' incisions that experienced an infection (superficial or deep) occurring up to and 21 days postoperatively between incisions treated with PICO compared with standard care dressings.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
participants
  PICO treatment with wound infection: number analyzed (Participants) | 197
  PICO treatment with wound infection | 4
  PICO treatment without wound infection: number analyzed (Participants) | 197
  PICO treatment without wound infection | 193
  Standard care with wound infection: number analyzed (Participants) | 197
  Standard care with wound infection | 6
  Standard care without wound infection: number analyzed (Participants) | 197
  Standard care without wound infection | 191

4. Secondary Outcome: Number of Participants Experiencing Postsurgical Incision Healing Complications (Delayed Healing) Occurring Within 7 Days Postoperatively
Description: Assessment of the number of participants' incisions that experienced delayed healing within 7 days of surgery between incisions treated with PICO compared with standard care dressings.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: Within 7 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery.
Measure: Number; unit: participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
participants
  PICO treatment with delayed healing | 102
  PICO treatment without delayed healing | 97
  Standard care with delayed healing | 103
  Standard care without delayed healing | 96

5. Secondary Outcome: Number of Participants Experiencing Postsurgical Incision Healing Complications (Delayed Healing) Occurring Within 10 Days Postoperatively
Description: Assessment of the number of participants' incisions that experienced delayed healing within 10 days of surgery between incisions treated with PICO compared with standard care dressings.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: Within 10 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery.
Measure: Number; unit: participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
participants
  PICO treatment with delayed healing | 64
  PICO treatment without delayed healing | 135
  Standard care with delayed healing | 64
  Standard care without delayed healing | 135

6. Secondary Outcome: Aesthetic Appearance (Cosmesis) and Scar Quality at 90 Days Postoperatively
Description: Assessment of the Patient and Observer Scar Assessment Scale (POSAS) and the Visual Analogue Scale (VAS) between postsurgical incisions treated with PICO compared with standard care dressings.
  VAS score: Assessed for color, appearance, contour, distortion, and texture. Each score ranged from 5 to 18; 5 being 'excellent' and 18 being 'poor.' Also, a global scar score was included in the total score.
  POSAS score: Scored in 2 parts which added to create a total score, observer score and patient score. The lowest score of 1 showed 'normal' skin and the highest score of 10 showed the 'worst imaginable' result.
  Observer score = 6 categories (vascularity, pigmentation, thickness, relief, pliability, and surface area) each given a score of 1-10.
  Patient score = 6 categories (scar pain, itching, color, stiffness, thickness, and irregularity each given a score of 1-10.
  All participants received both PICO and standard care dressings simultaneously during the course of the study.
Time Frame: 90 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery. All available results at the 90 day time point.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
score on a scale
  PICO - VAS Global Assessment: number analyzed (Participants) | 171
  PICO - VAS Global Assessment | 3 [1 to 9]
  Standard care - VAS Global Assessment: number analyzed (Participants) | 169
  Standard care - VAS Global Assessment | 3 [1 to 8]
  PICO - POSAS Observer Total: number analyzed (Participants) | 164
  PICO - POSAS Observer Total | 16 [7 to 41]
  Standard care - POSAS Observer Total: number analyzed (Participants) | 157
  Standard care - POSAS Observer Total | 18 [9 to 44]
  PICO - POSAS Patient Total: number analyzed (Participants) | 167
  PICO - POSAS Patient Total | 15 [6 to 51]
  Standard care - POSAS Patient Total: number analyzed (Participants) | 159
  Standard care - POSAS Patient Total | 19 [6 to 50]

7. Secondary Outcome: Number of Skin, Nipple and Areola Necrosis Occurring up to and 21 Days Postoperatively
Description: The nipple and areola areas were not covered by the PICO or standard care dressing as part of the evaluation, they were all dressed the same with Steri-strips and dry gauze pads, which was essentially the standard care dressing regime.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: There were 200 participants enrolled with 1 participant lost to follow-up immediately after surgery. All available results for this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
Participants
  PICO - skin necrosis: number analyzed (Participants) | 197
  PICO - skin necrosis | 2
  Standard care - skin necrosis: number analyzed (Participants) | 197
  Standard care - skin necrosis | 7
  PICO - nipple and areola necrosis: number analyzed (Participants) | 197
  PICO - nipple and areola necrosis | 2
  Standard care - nipple and areola necrosis: number analyzed (Participants) | 197
  Standard care - nipple and areola necrosis | 1

8. Secondary Outcome: Number of Hematoma's Occurring up to and 21 Days Postoperatively
Description: Assessment of participants developing a hematoma up to 21 days postoperatively for incisions treated with PICO compared with standard care dressings.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
Participants
  PICO - hematoma occurred: number analyzed (Participants) | 197
  PICO - hematoma occurred | 2
  Standard care - hematoma occurred: number analyzed (Participants) | 197
  Standard care - hematoma occurred | 3

9. Secondary Outcome: Number of Wounds Showing 100% Closure Occurring up to and 21 Days Postoperatively
Description: Assessment of wound appearance demonstrating 100% wound closure at 21 days postoperatively for both PICO treatment and standard of care treatment.
  All participants received both PICO and standard care dressings simultaneously during the course of the study; randomized to either right breast for PICO and left breast for standard of care OR right breast standard of care and left breast PICO.
Time Frame: 21 days postoperatively
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | PICO Negative Pressure Wound Therapy/Standard of Care Dressing
Number analyzed (Participants) | 199
Participants
  PICO - 100% wound closure: number analyzed (Participants) | 185
  PICO - 100% wound closure | 155
  Standard care - 100% wound closure: number analyzed (Participants) | 185
  Standard care - 100% wound closure | 134

ADVERSE EVENTS:
Time Frame: Baseline through 90 days postoperatively.
Groups:
- Standard of Care Dressing Arm: Adhesive Skin Closure Strips, e.g. STERI-Strips, or alternatively a non-adherent dry dressing if Adhesive Skin Closure Strips was not deemed appropriate by the Principle Investigator at that center.
Arm/Group | PICO Negative Pressure Wound Therapy | Standard of Care Dressing Arm
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 2/200 | 7/200
Other Adverse Events (participants affected / at risk) | 50/200 | 70/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICO Negative Pressure Wound Therapy (N=200) | Standard of Care Dressing Arm (N=200)
Epidermolysis at T-junction/skin trifurcation point (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Fat necrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 4 (4)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Infection and dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Severe postoperative pain (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PICO Negative Pressure Wound Therapy (N=200) | Standard of Care Dressing Arm (N=200)
Delayed wound healing (Skin and subcutaneous tissue disorders) | 50 (50) | 70 (70)

LIMITATIONS AND CAVEATS:
There was one site (68 enrolled participants in total) in which the data were analyzed separately due to issues at the site. This data was also analyzed and included in the overall totals for baseline characteristics and outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days